CLINICAL TRIAL: NCT02666456
Title: DOLORisk: Understanding Risk Factors and Determinants for Neuropathic Pain - The Influence of Sensory Phenotype on the Risk of Developing Neuropathic Pain
Brief Title: The Influence of Sensory Phenotype on the Risk of Developing Neuropathic Pain
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Kiel (Other)
Responsible Party: Principal Investigator, Andras Binder, PD Dr. med., University of Kiel
Other Study IDs: DOLORisk WP4
Record Dates: First submitted 2016-01-11; First posted 2016-01-28 (Estimated); Last update posted 2016-01-28 (Estimated); Status verified 2016-01

CONDITIONS: Neuropathic Pain; Polyneuropathy; Peripheral Nerve Injury
MeSH Terms: conditions — Neuralgia; Polyneuropathies; Peripheral Nerve Injuries | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cross-sectional cohort: Patients with chronic peripheral neuropathic pain
  Interventions: Other: QST, Questionnaires
- Longitudinal cohort: Painless patients before and after potential chronic neuropathic pain-inducing interventions (chemotherapy, Operation)
  Interventions: Other: QST, Questionnaires

INTERVENTIONS:
Other: QST, Questionnaires — Assessment of sensory phenotype by QST and questionnaires

SUMMARY:
Cross-sectional and longitudinal analysis of the somatosensory phenotype, assessed by quantitative sensory testing (QST) and Information obtained by questionnaires to detect risk factors for neuropathic pain development and chronification in painless and chronic pain patients.

ELIGIBILITY:
Inclusion Criteria:

* Chronic peripheral neuropathic pain or
* Painless Patient with risk to develop neuropathic pain (post-surgery, chemotherapy-induced)

Exclusion Criteria:

* Minors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Painless patients and patients with chronic peripheral neuropathic pain.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2016-04; Primary Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Somatosensory phenotype detected by quantitative sensory testing (QST) | Single assessment at baseline (cross-sectional study). Report of complete cohort data at study completion
  The somatosensory phenotype will be assessed by quantitative sensory testing (QST) once at baseline
Change of neuropathic pain: Development and chronification of neuropathic pain detected by DN4 questionnaire | Assessment of change of neuropathic pain from baseline and 6 months after study enrollment (longitudinal study). Report of complete cohort data at study completion.
  Assessment with DN4 pain questionnaire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Funding source — http://cordis.europa.eu/project/rcn/193238_en.html
- See also: WEbsite — http://www.ndcn.ox.ac.uk/research/neural-injury-group/research-projects/dolorisk